CLINICAL TRIAL: NCT04636463
Title: Music in Wide Awake Local Anesthesia no Tourniquet (WALANT) Hand Surgery: Prospective Randomized Control Trial
Brief Title: Music in Wide Awake Hand Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AILY20D.1059
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Hand Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Surgery with Music (Experimental): Participant undergoes surgery hand surgery using Wide Awake Local Anesthesia with no tourniquet (WALANT) while listing to music
  Interventions: Procedure: Intraoperative Music
- Hand Surgery without Music (Control Group) (No Intervention): Participant undergoes surgery hand surgery using Wide Awake Local Anesthesia with no tourniquet (WALANT) without listening to music

INTERVENTIONS:
Procedure: Intraoperative Music — Hand Surgery performed with the participant awake, using local anesthesia. Headphones will be worn by the participant and surgery will be performed while the participant is listening to music
  Arms: Hand Surgery with Music

SUMMARY:
Wide awake local anesthesia no tourniquet (WALANT) surgery has emerged as a popular technique in hand surgery over the last decade. It is possible that the unfamiliar sounds of the operating room could contribute to intraoperative patient anxiety during WALANT surgery. This study intends to investigate whether utilizing noise cancelling headphones and listening to music intraoperatively during WALANT hand surgery has an effect on patient anxiety, pain, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Already chose to undergo WALANT hand surgery with the participating surgeon

Exclusion Criteria:

- Age <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient anxiety levels will be recorded on a 10 point VAS scale | 3 hours
  Participant Satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States